CLINICAL TRIAL: NCT03012438
Title: The Use of Near-Infrared Fluorescence Imaging in Parathyroid Visualization During Thyroid Surgery: a Pilot Study
Brief Title: NIRF for Parathyroid Visualization: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL57409.068.16
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2017-04

CONDITIONS: Thyroid Disease
Keywords: Near infrared fluorescence; ICG; Parathyroid gland
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NIRF imaging in thyroid surgery (Experimental): 7.5 mg ICG is administered i.v. and the system will be switched to fluorescence mode. If needed, a second dose of 7.5 mg ICG can be administered. After identification of the parathyroid glands, surgery will continue until there is a desire to visualize the parathyroid glands again, another dose of ICG can be given. After complete removal of thyroid, another 7.5 mg of ICG will be given to assess the perfusion of the parathyroid gland. Directly after the procedure the researcher will ask the surgeon whether he/she thinks the technique is feasible.
  After surgery, the serum calcium levels will be determined in patients after total thyroidectomy on day 1, 2 and after two weeks. TSH will be determined after 2 weeks. The thyroid specimen will be send to pathology. In the specimen, the pathologist will search for parathyroid glands. Video recordings will be analyzed, quantifying the fluorescence signal compared to the background: measuring the TBR.
  Interventions: Device: NIRF imaging in thyroid surgery

INTERVENTIONS:
Device: NIRF imaging in thyroid surgery — a fluorescence imaging system and 7.5 mg of ICG will be used to visualize the parathyroids glands.
  Other Names: Near Infrared Fluorescence Imaging; Indocyanine green

SUMMARY:
During surgery in which the thyroid is removed (thyroidectomy), the identification of parathyroid glands, that should be saved, can be challenging. Therefore, there is need for accurate intraoperative guidance. Earlier animal studies show that the parathyroid glands can be identified by the use of the Near Infrared Fluorescent dye Indocyanine green (ICG).

Our hypothesis is therefore, that the use of ICG-based fluorescence imaging during thyroid surgery will provide real-time intraoperative visualization of the parathyroid glands.

This prospective observational feasibility study aims to evaluate the feasibility of the use of ICG in identifying the parathyroid glands during thyroid surgery. 30 patients (age >18 years) who are already regularly scheduled for thyroid surgery; i.e. patients undergoing total thyroidectomy are suitable for inclusion. In all patients, undergoing total thyroidectomy infrared fluorescence imaging, using a per-operative intravenous injection of 7.5 mg ICG, will be tested on feasibility and imaging characteristics.

DETAILED DESCRIPTION:
In this study, the feasibility of the use of NIR fluorescence imaging for the identification of the parathyroid glands during thyroid surgery will be explored.

Per-operatively: The surgery will start as usual. When the surgeon would normally search for the parathyroid glands, 7.5 mg of ICG will be administered intravenously through the infusion in the patients arm. An intravenous administration is chosen because of the minimal invasive nature and results of the described earlier case series in which ICG was also administered via peripheral infusion. Directly after that, the fluorescence system can be switched to fluorescence mode. The surgeon will determine whether the parathyroid glands are visible now. If needed, due to washout, a second dose of 7.5 mg of ICG can be administered. After identification of the parathyroid glands, surgery will continue as in the standard situation, until there is a desire to visualize the parathyroid glands again, then another dose of ICG can be given. Time until first identification of the parathyroid glands and total surgical time will be measured. After complete removal of the thyroid, another 7.5 mg of ICG will be administered intravenously to visualize the vascularization of the parathyroid gland. The intensity will be subjectively scored: 1 parathyroid black after injection of ICG, 2 partially vascularized, or 3 parathyroid is green; well vascularized. The fluorescence system will be used to record the whole procedure. Directly after the procedure the researcher will ask the surgeon whether he or she thinks the technique is feasible.

Postoperatively: As in standard care, after thyroid surgery, the serum calcium levels will be determined. Low calcium levels can indicate misidentification of parathyroid glands. These calcium levels are determined only in patients after total thyroidectomy on day 1, 2 and after two weeks. Also TSH will be determined after two weeks as in standard care. The thyroid specimen will be send to pathology. In the specimen, the pathologist will search for parathyroid glands, as is standard care. Furthermore, video recordings will be analyzed, quantifying the fluorescence signal compared to the background: measuring the Target to Background Ratio. Also, in these video recordings the time until visualization of the parathyroid glands will be reassessed by an independent expert.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged 18 years and above
* Scheduled for elective total or hemi thyroidectomy
* Normal liver and renal function
* No known hypersensitivity for iodine or ICG
* Able to understand the nature of the study procedures
* Willing to participate and give written informed consent

Exclusion Criteria:

* Age < 18 years
* Liver or renal insufficiency
* Known ICG, iodine, penicillin or sulfa hypersensitivity
* Pregnancy or breastfeeding
* Not able to understand the nature of the study procedure
* i.v. heparin injection in the last 24h (LMWH not contraindicated)
* Not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Time to identification of parathyroid glans | during surgery
  Can the parathyroid glands be identified earlier with NIRF light? Time until identification in NIRF and white light will be compared.

SECONDARY OUTCOMES:
Total surgical time | From incision until closure
Histology: are parathyroid glands in the specimen? (as in standard care) | assessment within 1 week after surgery
  immediately after surgery, the thyroid specimen will be send to the pathology department for histological examination as in standard care, with extra attention on wether there are parathyroid glands in the specimen.
Subjective opinion surgeon about the usefulness of the technique | Immediately after surgery
Intra-operative complications due to the use of the technique | during surgery

OTHER OUTCOMES:
Quantitative measurement of fluorescence signal related to parathyroid function | up to 2 weeks
  Quantitative measurement of fluorescence signal using Target to Background Ratio (TBR) is used, combined with parameters of parathyroid function, namely Calcium levels postoperatively day 1 and day 2, and week 2 in patients after total thyroidectomy (as in standard care), and TSH in patients after total thyroidectomy 2 weeks postoperatively (as in standard care).

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Bouvy, M.D. Ph.D., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No